CLINICAL TRIAL: NCT01903005
Title: A Multi-center, Open-Label, 24-Week, Follow-Up Study to Assess Safety, Efficacy, and Treatment Adherence For Maintenance Treatment of Opioid Dependence With OX219
Brief Title: Multi-Center, Open-Label, 24-Week Study of OX219 Safety and Efficacy for Maintenance Treatment of Opioid Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orexo AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX219-008
Record Dates: First submitted 2013-07-09; First posted 2013-07-19 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Opioid Dependence, on Agonist Therapy
Keywords: Opioid, Dependence, agonist, Buprenorphine, Naloxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label BNX sublingual tablets (Experimental): Weeks 1-24: Higher bioavailability BNX sublingual tablets (open-label) were titrated at doses ranging from 5.7/1.4 mg to 17.1/4.2 mg, to a dose that relieved opioid cravings and withdrawal symptoms with minimal side effects.
  Interventions: Drug: Higher bioavailability BNX sublingual tablets

INTERVENTIONS:
Drug: Higher bioavailability BNX sublingual tablets — Once daily, open-label treatment with higher bioavailability BNX sublingual tablets for 24 weeks
  Other Names: OX219; Zubsolv; Buprenorphine/naloxone sublingual tablets

SUMMARY:
The purpose of this study was to assess safety, efficacy, and treatment retention following extended treatment with OX219, a higher-bioavailability buprenorphine/naloxone (BNX) sublingual tablet formulation in opioid-dependent patients who completed 1 of 2 primary efficacy and safety studies of OX219.

DETAILED DESCRIPTION:
This was a multicenter, open-label, uncontrolled, single-arm, 24-week, extension study to assess safety, efficacy, and treatment retention during maintenance treatment.

Eligible patients had completed 1 of 2 primary efficacy and safety studies of the higher-bioavailability BNX sublingual tablet formulation (primary study OX219-006 [NCT01908842] or OX219-007 [NCT01848054]). The total duration of study treatment was 24 weeks.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent form.
* Completion of 1 of 2 primary efficacy safety studies of BNX sublingual tablets (OX219-006 or OX219-007).
* Female patients of child bearing potential who used a reliable method of contraception (hormonal, condom with spermicide, intrauterine device) during the previous OX219-006 or OX219-007 study and continue to use it for the OX219-008 study. Females who are not of child-bearing potential who are either surgically sterile (by hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or tubal ligation), or postmenopausal, as defined by being at least 50 years of age and having had an absence of menses for at least 2 years, were also eligible.

Exclusion criteria

* Females who are pregnant (positive pregnancy test result) or lactating, or planning to become pregnant during the study.
* Participants who are unwilling or unable to comply with the requirements of the protocol (eg, pending incarceration) or are in a situation or condition that, in the opinion of the investigator, may interfere with participation in the study.
* Participants who are participating in any other clinical study in which medication(s) are being delivered or who had used an investigational drug or device within the last 30 days.
* Participants with any known allergy or sensitivity or intolerance to buprenorphine, naloxone, or any related drug, or history of any drug hypersensitivity or intolerance that, in the opinion of the investigator, would compromise the safety of the subject or the study.
* Participant with a contra-indicated serious medical condition.
* Participants who are at suicidal risk as determined by any of the following: a history of suicidal ideation ≤ 3 months prior to baseline with a score of 4 (intent to act) or 5 (specified plan and intent) on the Columbia Suicide Severity Risk Scale (C-SSRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hoffman, Principal Investigator — TRY Research, 406 Lake Howell Road, Maitland, Florida 32751
Locations (28):
- United States (28):
  - Jefferson County, Alabama
  - Marion County, Alabama
  - Winston County, Alabama
  - Maricopa County, Arizona
  - Los Angeles County, California
  - San Diego County, California
  - Broward County, Florida
  - Columbia County, Florida
  - Duval County, Florida
  - Jacksonville Metropolitan Area, Florida
  - Miami-Dade County, Florida
  - Orlando Metropolitan Area, Florida
  - Osceola County, Florida
  - Palm Beach County, Florida
  - DeKalb County, Georgia
  - Chicago Metropolitan Area, Illinois
  - Baltimore County, Maryland
  - Bristol County, Massachusetts
  - Rankin County, Mississippi
  - Saint Louis Metropolitan Area, Missouri
  - Warren County, New Jersey
  - Oklahoma County, Oklahoma
  - Portland Metropolitan Area, Oregon
  - Delaware County, Pennsylvania
  - Philadelphia County, Pennsylvania
  - Charleston County, South Carolina
  - Salt Lake County, Utah
  - Benton County, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 668 patients who completed primary study OX219-006 (NCT01908842) or OX219-007 (NCT01848054) were enrolled. Three patients entered the study without taking any study medication and were excluded. A total of 665 patients were included in the data analyses.
Groups:
- Safety Population: Weeks 1-24: Higher bioavailability BNX sublingual tablets (open-label) were titrated at doses ranging from 5.7/1.4 mg to 17.1/4.2 mg, to a dose that relieved opioid cravings and withdrawal symptoms with minimal side effects.
Period: Overall Study
Arm/Group | Safety Population
Started | 665 (Primary study OX219-006 (n=475); Primary study OX219-007 (n=190))
Completed | 292 (Primary study OX219-006 (n=194); Primary study OX219-007 (n=98))
Not Completed | 373

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- OX219-006 Completers; OX219-007 Completers: Weeks 1-24: Higher bioavailability BNX sublingual tablets (open-label) were titrated at doses ranging from 5.7/1.4 mg and 17.1/4.2 mg, to a dose that relieved opioid cravings and withdrawal symptoms with minimal side effects.
- Total: Total of all reporting groups
Arm/Group | OX219-006 Completers | OX219-007 Completers | Total
Number analyzed (Participants) | 475 | 190 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.4) | 39.0 (10.8) | 36.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 63 | 259
  Male | 279 | 127 | 406
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 17 | 82
  Not Hispanic or Latino | 410 | 173 | 583
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 21 | 83
  White | 402 | 167 | 569
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 5 | 0 | 5
Height [Mean (Standard Deviation); unit: cm] | 171.99 (9.43) | 173.35 (10.01) | 172.38 (9.61)
Weight [Mean (Standard Deviation); unit: kg] | 78.34 (18.99) | 78.98 (20.73) | 78.53 (19.49)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.47 (6.11) | 26.26 (6.63) | 26.41 (6.26)
Duration of Opioid Use [Median (Standard Deviation); unit: years] | 7.20 (9.50) | 9.6 (8.79) | 7.95 (9.32)

OUTCOME MEASURES:

1. Secondary Outcome: Retention in Treatment in the Safety Population
Description: Retention in treatment by visit in the safety population at weeks 4, 8, 12, 16, 20, and 24, defined as the number of patients receiving treatment on the day of the visit (± 5 days for each visit)
Time Frame: Treatment retention was assessed at weeks 4, 8, 12, 16, 20, and 24
Population: Safety population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 665
participants
  Week 4 | 563 [545 to 581]
  Week 8 | 483 [460 to 505]
  Week 12 | 425 [401 to 450]
  Week 16 | 383 [358 to 408]
  Week 20 | 333 [308 to 358]
  Week 24 | 292 [267 to 317]

2. Secondary Outcome: Mean Change From Primary Study Baseline (OX219-006 or OX219-007) in Clinical Opioid Withdrawal Scale (COWS) Score
Description: Mean change from primary study baseline in COWS total scores during the 24-week open-label, extension study; COWS scores range from 0 to 48, with a lower score being more favorable; study endpoint was defined as the last post-baseline value recorded for COWS
Time Frame: Prior to dosing on day 1, at weeks 4, 8,12,16, 20, 24, and at study endpoint
Population: Safety population; patient population at day 1 (n=658) is lower than overall safety population (n=665) due to missing data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Safety Population
Number analyzed (Participants) | 665
units on a scale
  Day 1 (n=658) | -12.0 [-12.3 to -11.6]
  Week 4 (n=557) | -12.2 [-12.6 to -11.8]
  Week 8 (n=477) | -12.7 [-13.1 to -12.3]
  Week 12 (n=423) | -12.9 [-13.4 to -12.5]
  Week 16 (n=384) | -13.1 [-13.6 to -12.6]
  Week 20 (n=336) | -13.3 [-13.8 to -12.8]
  Week 24 (completers only; n=288) | -13.1 [-13.7 to -12.6]
  Study Endpoint (n=597) | -12.5 [-12.9 to -12.1]

3. Secondary Outcome: Mean Change From Primary Study Baseline (OX219-006 or OX219-007) in Subjective Opioid Withdrawal Scale (SOWS) Score
Description: Mean change from primary study baseline in SOWS total scores during the 24-week open-label, extension study; SOWS scores range from 0 to 64, with a lower score being more favorable; study endpoint was defined as the last post-baseline value recorded for SOWS
Time Frame: Prior to dosing on day 1, at weeks 4, 8,12,16, 20, and 24, and at study endpoint
Population: Safety population; patient population at day 1 (n=650) is lower than overall safety population (n=665) due to missing data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Safety Population
Number analyzed (Participants) | 665
units on a scale
  Day 1 (n=650) | -26.8 [-27.8 to -25.7]
  Week 4 (n=550) | -27.4 [-28.6 to -26.2]
  Week 8 (n=472) | -28.0 [-29.2 to -26.7]
  Week 12 (n=418) | -27.7 [-29.0 to -26.3]
  Week 16 (n=376) | -28.7 [-30.1 to -27.3]
  Week 20 (n=331) | -28.9 [-30.4 to -27.5]
  Week 24 (n=282) | -27.7 [-29.4 to -26.0]
  Study Endpoint (n=588) | -27.3 [-28.5 to -26.1]

4. Secondary Outcome: Mean Change From Primary Study Baseline (OX219-006 and OX219-007) in Visual Analog Scale (VAS) Craving Scores
Description: Mean change from primary study baseline in VAS craving scores during the 24-week open-label, extension study; VAS craving scores range from 0 ("no cravings") to 100 mm ("most intense craving I have ever had"); study endpoint was defined as the last post-baseline value recorded for VAS craving
Time Frame: Prior to dosing on day 1, at weeks 4, 8, 12, 16, 20, and 24, and at study endpoint
Population: Safety population; patient population at day 1 (n=646) is lower than overall safety population (n=665) due to missing data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Safety Population: Weeks 1-24: Higher bioavailability BNX sublingual tablets (open-label) were titrated at doses ranging 5.7/1.4 mg to 17.1/4.2 mg, to a dose that relieved opioid cravings and withdrawal symptoms with minimal side effects.
Arm/Group | Safety Population
Number analyzed (Participants) | 665
units on a scale
  Day 1 (n=646) | -52.8 [-55.0 to -50.6]
  Week 4 (n=563) | -56.6 [-59.0 to -54.2]
  Week 8 (n=479) | -59.4 [-62.0 to -56.9]
  Week 12 (n=426) | -59.4 [-62.0 to -56.8]
  Week 16 (n=384) | -61.5 [-64.1 to -58.8]
  Week 20 (n=338) | -61.4 [-64.3 to -58.5]
  Week 24 (n=289) | -60.5 [-63.8 to -57.2]
  Study Endpoint (n=598) | -57.3 [-59.6 to -55.0]

5. Secondary Outcome: Percent Change From Primary Study Baseline (OX219-006 or OX219-007) for Question 1 of the Work Productivity/Activity Impairment: 6-Question Specific Health Problem Questionnaire (WPAI:SHP)
Description: Question 1 of the WPAI:SHP asks patients to provide a "yes" or "no" response to the question "Are you employed?"; The percentage of patients employed at the end of the 24-week open-label, extension study was calculated by subtracting the percentage of previously employed patients not employed at study end from the percentage of previously unemployed patients who were employed by study end
Time Frame: Study Endpoint
Population: Safety population; patients with missing data were excluded from the analysis and are reflected in the number of patients analyzed
Measure: Number; unit: percentage of patients
Arm/Group | Safety Population
Number analyzed (Participants) | 665
percentage of patients
  Unemployed at baseline; employed at study endpoint | 21.3
  Employed at baseline; unemployed at study endpoint | 6.0
  Increase in patients employed at study endpoint | 15.3

6. Secondary Outcome: Mean Change From Primary Study Baseline (OX219-006 or OX219-007) for Questions 2-4 of the WPAI:SHP
Description: Mean change from primary study baseline to week 24 of the open-label, extension study for questions 2-4 of the WPAI:SHP; Question 2: During the past 7 days, how many hours did you miss from work because of problems associated with your opioid dependence?; Question 3: During the past 7 days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study?; Question 4: During the past 7 days, how many hours did you actually work?
Time Frame: Week 24
Population: Safety population; patients with missing data were excluded from the analysis and are reflected in the number of participants analyzed
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Safety Population
Number analyzed (Participants) | 665
hours
  Missed work hours due to opioid dependence (n=79) | -4.8 [-8.1 to -1.5]
  Missed work hours due to other reason (n=79) | -0.2 [-1.9 to 1.5]
  Number of hours actually worked (n=78) | 7.7 [3.4 to 12.0]

7. Secondary Outcome: Mean Change From Primary Study Baseline (OX219-006 or OX219-007) for Questions 5-6 of the WPAI:SHP
Description: Mean change from primary study baseline to week 24 of the open-label extension study for questions 5-6 of the WPAI:SHP; Question 5: During the past 7 days, how much did your opioid dependence affect your productivity while you were working?; Question 6: During the past 7 days, how much did your opioid dependence affect your ability to do regular daily activities, other than work at a job?; Questions 5 and 6 of the WPAI:SHP are scored on an 11-point scale (0 = problem had no effect; 10 = problem completely prevented me from doing my work/daily activities)
Time Frame: Week 24
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Safety Population
Number analyzed (Participants) | 665
units on a scale
  Problem affects work productivity (n=70) | -3.9 [-4.7 to -3.1]
  Problem affects daily activities (n=283) | -4.3 [-4.8 to -3.9]

8. Primary Outcome: Number of Patients Reporting Treatment-Emergent Adverse Events
Description: Number of patients reporting treatment-emergent adverse events during open-label, extension treatment with higher bioavailability BNX sublingual tablets
Time Frame: Day 1 through week 24
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 665
participants
  Constipation | 20
  Headache | 21

9. Primary Outcome: Number of Patients Reporting Treatment-Related, Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events considered related to treatment with the higher bioavailability BNX sublingual tablets
Time Frame: Day 1 through week 24
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 665
participants
  Gastrointestinal disorders | 32
  Constipation | 19

10. Primary Outcome: Number of Patients Reporting Treatment-Emergent Serious Adverse Events
Description: Patients reporting treatment-emergent serious adverse events considered either related or not related to treatment with the higher bioavailability BNX sublingual tablets
Time Frame: Day 1 throught week 24
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 665
participants
  Possibly treatment-related | 1
  Not treatment-related | 8

11. Primary Outcome: Number of Patient Discontinuations Due to Treatment-Emergent Adverse Events
Description: Study discontinuations due to treatment-emergent adverse events that occurred during treatment with bioavailability BNX sublingual tablets
Time Frame: Day 1 through week 24
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 665
participants | 14

ADVERSE EVENTS:
Time Frame: Day 1 through Week 24 of Open-Label Extension Study
Description: Safety population (N=665)
Groups:
- Safety Population: Weeks 1-24: Higher bioavailability BNX sublingual tablets (open-label) were titrated at doses of buprenorphine/naloxone between 5.7/1.4 mg and 17.1/4.2 mg mg, to a dose that relieved opioid cravings and withdrawal symptoms with minimal side effects.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 15/665
Other Adverse Events (participants affected / at risk) | 41/665
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=665)
Heroin toxicity (Injury, poisoning and procedural complications) | 1 (1) — Condition led to death; non-treatment-emergent; not related to study drug.
Hypertensive and atherosclerotic cardiovascular disease (Cardiac disorders) | 1 (1) — Condition led to death; non-treatment-emergent, not related to study drug.
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Moderate, treatment-emergent; not related to study drug.
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) — Moderate, treatment-emergent; not related to study drug.
Depression (Psychiatric disorders) | 2 (2) — Mild, treatment-emergent; not related to study drug in one patient; severe, treatment-emergent; possibly related to study drug in another patient.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Moderate, treatment-emergent; not related to study drug.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Moderate, treatment-emergent; not related to study drug.
Anal abscess (Infections and infestations) | 1 (1) — Severe, treatment-emergent; unlikely related to study drug.
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) — Moderate, treatment-emergent; not related to study drug.
Overdose (Injury, poisoning and procedural complications) | 1 (1) — Severe, treatment-emergent; not related to study drug.
Metabolic encephalopathy (Nervous system disorders) | 1 (1) — Severe, treatment-emergent; not related to study drug.
Urinary tract infection (Infections and infestations) | 1 (1) — Severe, treatment-emergent; not related to study drug.
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) — Severe, treatment-emergent; not related to study drug.
Intentional overdose (Social circumstances) | 1 (1) — Severe, non-treatment-emergent; not related to study drug.
Worsening of opioid dependence (Psychiatric disorders) | 2 (2) — Moderate, non-treatment-emergent; not related to study drug in two patients.
Bipolar depression (Psychiatric disorders) | 1 (1) — Severe, non-treatment-emergent; unlikely related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=665)
Constipation (Gastrointestinal disorders) | 20 (22) — Treatment-emergent.
Headache (Nervous system disorders) | 21 (22) — Treatment-emergent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No